CLINICAL TRIAL: NCT06130098
Title: Investıgatıon Of The Effect Of Traınıng And Counselıng Provıded By Tele Nursıng Servıce After Total Knee Prosthesıs On Post-Operatıve Qualıty Of Lıfe And Complıcatıons
Brief Title: Investıgatıon Of The Effect Of Traınıng And Counselıng Provıded By Tele Nursing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, GÜLŞAH BEKTAŞ, LECTURER, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HasanKU-HEM-GB-01
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Musculoskeletal Diseases
Keywords: total knee replacement; telenursing; post-discharge care
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: There are two groups: control and study groups. Certain applications were planned to be applied to the control group and the study group.
Who Masked: Participant, Investigator
Masking Description: Randomized: Participants are assigned to intervention groups by chance and control groups will be established. In the randomization method, whether the participants will be in the study group or the control group will be determined by the simple random numbers method using a computer program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Training by the clinical nurse before discharge. Prepare an educational brochure and give it to patients. Application of patient information form, EQ-5D-5L Quality of Life and Oxford Knee Score Scale During the routine check-up in the first week, evaluates the development of complications without knowing which group the patient is in.
  Within the first week and at the end of the fourth week, the wound site is evaluated by the physician for the development of complications, . Patients who cannot come for a check-up should send a photo of the wound area to the researcher via WhatsApp application, and the photo will be forwarded to the clinician who performed the surgery and the physician will record the complication situation. It is planned to receive complication development and wound site evaluation results from the physician system.
  At the end of the fourth and sixth weeks after discharge, the EQ-5D-5L and OKS scale must be filled in again by the patients.
  Interventions: Other: control group
- experimental group (Active Comparator): Active Comparator: experimental group Providing education to patients by preparing a pre-discharge education brochure. You will be contacted by phone at the end of the first, second, third and fourth weeks after discharge.
  Application of the patient information form, EQ-5D-5L Quality of Life and Oxford Knee Score Scale. Evaluation of the wound site in terms of complications at the end of the first and fourth weeks. It is planned to receive complication development and wound site evaluation results from the system.
  After the first check-up, a call is made at the end of the first week after discharge.
  Providing training on the subjects included in the training brochure during the first phone call
  In the fourth meeting, tele-nursing service was provided through the "Telephone Counseling Protocol"
  Refilling of the EQ-5D-5L quality of life and Oxford Knee Score scale by patients at routine check-up at the end of the fourth and sixth weeks after discharge
  Interventions: Other: experimental group

INTERVENTIONS:
Other: control group — Training by the clinical nurse before discharge. Prepare an educational brochure and give it to patients. Application of patient information form, EQ-5D-5L Quality of Life and OKS Scale During the routine check-up in the first week, evaluates the development of complications without knowing which group the patient is in.
  Within the first week and at the end of the fourth week, the wound site is evaluated by the physician for the development of complications, . Patients who cannot come for a check-up should send a photo of the wound area to the researcher via WhatsApp application, and the photo will be forwarded to the clinician who performed the surgery and the physician will record the complication situation. It is planned to receive complication development and wound site evaluation results from the physician system.
  At the end of the fourth and sixth weeks after discharge, the EQ-5D-5L and OKS scale must be filled in again by the patients.
  Arms: control group
Other: experimental group — Providing training before discharge Prepare an educational brochure and give it to patients. You will be contacted by phone at the end of the first, second, third and fourth weeks after discharge.
  Application of patient information form, EQ-5D-5L Quality of Life and OKS Scale Evaluating the wound site in terms of complications within the first week and at the end of the fourth week. It is planned to receive complication development and wound site evaluation results from the system.
  After the first check-up, calling the patients in the study group at the end of the first week after discharge.
  Providing training on the subjects included in the training brochure in the first phone call and recording any existing problems.
  In the fourth meeting, tele-nursing service will be provided through the "Telephone Counseling Protocol".
  EQ-5D-5L and OKS forms must be filled out again by patients at the routine check-up at the end of the fourth and sixth weeks after discharge.
  Arms: experimental group

SUMMARY:
To examine the effect of education and consultancy provided via telenursing service after total knee arthroplasty on postoperative quality of life and some complications.

DETAILED DESCRIPTION:
It is estimated that osteoarthritis, which causes low quality of life in old age and is one of the serious obstacles to physical independence, affects more than 250 million people in the world, as the elderly population in the world and in our country increases. Osteoarthritis is characterized by degeneration of joint cartilage, accompanied by pain and loss of function, and its etiology is not yet fully known; It is a chronic joint disease that is accompanied by metabolic, genetic and other affecting factors.

The most common area of osteoarthritis is the knees, and its progression is generally slow. Knee osteoarthritis is a public health problem due to increasing age, obesity and the increase in knee traumas. Knee osteoarthritis begins to occur at the age of 40 and is estimated to be more common in women than in men. According to World Health Organization (WHO) data, osteoarthritis is seen at a rate of 18% in women aged 60 and over and 9.6% in men (6). It has been stated that the prevalence of osteoarthritis increases as the elderly population increases in the USA, and 62% of osteoarthritis patients in New Zealand have knee osteoarthritis. According to the Health Survey data conducted by the Turkish Statistical Institute (TUIK) (2019) in our country, it is stated that 11.2% of the population has problems related to osteoarthritis.

Knee osteoarthritis is a disease with multiple etiologies consisting of regional and systemic factors. There are modifiable and non-modifiable risk factors such as age, gender, nutrition, genetics, obesity, trauma, alignment disorders, occupation, physical activity, and muscle weakness. In the treatment of knee osteoarthritis, total knee prosthesis (TKA) is applied to patients when conservative approaches such as medical and physical therapy are insufficient and surgical interventions such as osteotomy and debridement fail to yield results. TDP; It is the process of replacing the damaged joint surface (tibial, femoral, patellar joint surfaces) in the knee, which develops due to osteoarthritis, rheumatoid arthritis, post-traumatic arthritis and other nonspecific arthritis, with metal or polyethylene prostheses. The purpose of total knee prosthesis is; It is applied to increase knee joint functions, correct deformities, reduce pain, and also improve the quality of life of individuals.

Patients who undergo TKA surgery are generally in the elderly group. In this group, patients with chronic diseases (atherosclerotic heart disease, hypertension, diabetes mellitus, chronic obstructive lung), those who have previously undergone orthopedic surgery, long-term surgery, inappropriate prosthesis selection for the individual, metabolic problems, soft tissue problems, problems in bone tissue and prosthesis design. Errors in application technique increase the risk of morbidity and mortality before, during and after TKA surgery.

Since FFP surgery is a major orthopedic surgical intervention, it can lead to serious complications. These complications; Complications related to the wound site include neurovascular complications (deep vein thrombosis, pulmonary embolism), infection (superficial infection, deep infection), patellafemoral problems, instability, joint stiffness, early aseptic loosening, osteolysis and periprosthetic fracture formation. Especially in case of serious complications such as aseptic loosening, infection and pain, the patient cannot use the prosthesis and revision may be required.

Nurses working in the field of orthopedics have an important role in reducing/preventing complications and re-surgeries related to TKA surgery, increasing patient satisfaction and reducing care costs. Basic principles of orthopedic nursing in patients who will undergo TKA surgery; It includes preventing possible complications, ensuring the functionality of the knee and preserving mobilization. At the same time, orthopedic nurses should give detailed counseling to patients, starting from the preoperative period, about preoperative preparation, surgical procedure, postoperative care, home care after discharge (medication use, exercise, nutrition, wound care, etc.), complications that may develop and initiatives to prevent them. . The advisory role of the nursing profession; It is expected that the society will recognize and use its own opportunities and resources regarding protecting and improving public health, increasing the quality of life, coping with disease-related problems, and ensuring that patients have access to scientific information. Effective counseling carried out by the nurse; It accelerates recovery and facilitates the adaptation of the patient and his family to the process.

Today, patients are discharged early after surgery due to the insufficient number of beds in hospitals, the cost of long-term stays, and the increased risk of infection. Early discharge can turn into a troublesome process for the patient and his family. Because many patients cannot adequately prepare for the post-operative recovery period at home, they feel inadequate and insecure during this process, and their recovery period can last up to a month.

ELIGIBILITY:
Inclusion Criteria:

* Having TDP surgery for the first time,
* Having primary elective TKA surgery,
* Having had a single (unilateral) knee prosthesis surgery,
* Patients whose FFP indication is osteoarthritis,
* No hearing, understanding, vision or speaking problems,
* Agreeing to participate in the research voluntarily,
* Able to understand and speak Turkish,
* Least literate,
* Those who have a mobile phone that can take photos of themselves or those nearby,
* Patients who have a smartphone or a smartphone nearby,
* Patients who do not develop serious complications that will delay discharge from the hospital

Exclusion Criteria:

* Answering data collection forms incompletely
* Being illiterate in Turkish
* Patients who agreed to participate in the study but later left
* Patients who cannot be reached when called and whose follow-up cannot be completed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-11-13 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
OXFORD KNEE SCORE | at the end of the fourth and sixth weeks
  To evaluate the gains in daily life and the change in the health of patients who haveundergone TKA surgery after surgery.The scoring system is a 12-item self-reported measurement tool to evaluate physical function and pain in patients with total knee arthroplasty. After this scoring system is applied, the answers given by the patients are scored between 0 and 4. In total, a patient can get a minimum of 0 and a maximum of 48 points. For results, 0-19 points are considered excellent, 20-29 points are good, 30-39 points are fair, and 40-48 points are considered poor.

SECONDARY OUTCOMES:
EQ-5D-5L quality of life scale | at the end of the fourth and sixth weeks
  To evaluate the quality of life.It consists of two parts. The first part is the health profile of that day; It allows it to be defined in five sub-dimensions: movement, self-care, usual activities, pain / discomfort and anxiety / depression. Answers given in each section; It has 5 options: "no problem", "mild problem", "moderate problem", "severe problem" and "extreme problem". The second part consists of the visual analog scale (VAS). In this section, individuals give values between 0 and 100 about their current health status and mark it on a thermometer-like scale. Quality of life scores ranging from 0 to 100 are obtained from the visual analog scale section. As the score of the scale increases, the perception of health increases positively.

CONTACTS AND LOCATIONS:
Overall Officials: HasanKU HasanKU, LECTURER, Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Nevşehir Devlet Hastanesi, Nevşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No